CLINICAL TRIAL: NCT01347996
Title: Open-Label, Multicenter, Effects of Remission Maintenance Therapy With Ceplene® , Given in Conjunction With Low-Dose Interleukin-2, on Immune Response and Minimal Residual Disease in Adult Patients With AML in First Complete Remission
Brief Title: Maintenance Therapy With Ceplene® (Histamine) and IL-2 on Immune Response and MRD in Acute Myeloid Leukemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cytovia, Inc. (Other)
Collaborators: EpiCept Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPC2008-02
Record Dates: First submitted 2011-05-02; First posted 2011-05-05 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Leukemia; Acute Myeloid Leukemia; Minimal Residual Disease; Ceplene; Histamine; interleukin 2
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Neoplasm, Residual | interventions — Histamine; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- histamine dihydrochloride and IL-2 (Experimental): histamine and IL-2 subcutaneous injections
  Interventions: Drug: histamine dihydrochloride and IL-2

INTERVENTIONS:
Drug: histamine dihydrochloride and IL-2 — Ceplene 0.5 mg subcutaneously twice daily and IL-2 1 µg/kg [16,400 IU/kg] body weight twice daily for 10, 21 day cycles
  Other Names: Ceplene; Proleukin; IL-2; interleukin-2; histamine

SUMMARY:
Ceplene/IL-2 remission maintenance therapy has been shown to significantly prolong Leukemia Free Survival in patients with Acute Myeloid Leukemia (AML) in first complete remission. This is an international, multicenter, open-label study to evaluate the effects of remission maintenance therapy with Ceplene/IL-2 in adult patients with AML in CR1 on specific immune system cells (T and NK cells) and prospectively defined markers of immune response that are known to reflect T and NK cell ability to combat AML.

DETAILED DESCRIPTION:
Outcome Measures:

Primary:

1. To assess the quantitative and qualitative pharmacodynamic effects of Ceplene plus low-dose IL-2 (Ceplene/IL-2) by monitoring T and natural killer (NK) cell phenotypes and their functionality after the first and third treatment cycles in adult patients with acute myeloid leukemia (AML) in first complete remission (CR1).
2. To evaluate minimal residual disease (MRD) in AML patients receiving Ceplene/IL-2.

Secondary:

To document, in adult AML patients in CR1 treated with Ceplene/IL-2:

1. Leukemia-free survival (LFS) after a follow-up period of up to two years.
2. The safety of Ceplene/IL-2 therapy.
3. The potential relationship of Ceplene/IL-2 effects on T and NK cell phenotypes and their functionality to MRD.

ELIGIBILITY:
Inclusion Criteria:

* AML patients in CR1 whose AML subtype has been well-characterized using conventional karyotyping and molecular genetic techniques (eg, RQ-PCR) at diagnosis. Patients may be considered eligible if they have not had this assessment performed at diagnosis provided that stored samples of diagnostic genetic material (DNA/RNA) from blood and BM are available that can be assayed for the presence of markers such as WT1 and/or AML-specific genetic markers.
* Bone marrow examination confirming CR (defined as less than 5% blasts in a normocellular bone marrow).
* Eighteen years of age or older.
* Patients have received any form of induction and consolidation therapy as per standard practice at the institution, including autologous stem cell transplantation (ASCT).
* Within 8 weeks following the date of the last dose of consolidation or conditioning chemotherapy for AML, or following ASCT.
* Patients not undergoing consolidation therapy must have been in CR1 for at least one month prior to enrollment.
* Platelet count recovered after chemotherapy to ≥75 x 109/L, and Partial Thromboplastin Time (PTT) within normal limits.
* WBC ≥1.5 x 109/L and LFTs (to include SGPT [ALAT] or SGOT [AST] and bilirubin) should not exceed twice the upper limit of normal.
* Serum creatinine less than or equal to 1.5 times the upper normal limit.
* Able to function without significant decrease in daily activities (WHO Performance Status 0 - 1 or Karnofsky ≥70).
* Life expectancy of more than three months and able to undergo routine outpatient evaluations for efficacy, safety, and/or compliance.
* Women of childbearing potential must be practicing barrier or oral contraception, for the duration of the treatment, or documented as surgically sterile or one year post-menopausal.
* If female, be non-nursing, non-pregnant and have a negative pregnancy test within two weeks of starting study drug.
* The patient must be informed of the investigational nature of the study and written informed consent obtained.

Exclusion Criteria:

* Patients who have undergone or are planned for allogeneic stem cell transplantation.
* Patients with M3 as an AML subtype.
* Class III or IV cardiac disease, hypotension or severe hypertension, vasomotor instability, serious or uncontrolled cardiac dysrhythmias (including ventricular arrhythmias) at any time, acute myocardial infarction within the past 12 months, active uncontrolled angina pectoris or symptomatic arteriosclerotic blood vessel disease.
* Other active malignancies except in situ carcinoma of the cervix, localized squamous or basal cell carcinoma of the skin.
* Serious concurrent or recent non-malignant medical conditions which, in the opinion of the Investigator, makes the patient unsuitable for participation in this study.
* History of seizures, central nervous system disorders, stroke within the last 12 months, or psychiatric disability thought to be clinically significant in the opinion of the Investigator and adversely affecting compliance to protocol.
* Patients unable to undergo repeat treatments, clinical evaluations and other diagnostic procedures required by the protocol.
* Active autoimmune disease (including but not limited to systemic lupus, inflammatory bowel disease, and psoriasis).
* Patients with active peptic or esophageal ulcer disease or with past peptic ulcer or esophageal disease with a history or bleeding.
* Patients requiring active treatment for hypotension.
* Medical, sociologic, or psychological impediment to probable compliance with the protocol.
* Patients continuing systemic treatment with clonidine, steroids, and/or H2 receptor blocking agents.
* Patients with a history of histamine hypersensitivity, severe allergies to food or contrast media requiring treatment within the last five years.
* Patients unable to provide written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) in AML patients receiving Ceplene/IL-2 | Comparison at baseline and various time points up to 2 years
  A second primary objective of this study is to evaluate MRD in patients who are receiving remission maintenance therapy with Ceplene/IL-2. MRD will be evaluated using RQ-PCR for molecular detection of genetic markers of AML. Patients' MRD status will be quantified at the time of enrollment (baseline) and within ten days after completion of Cycles 3, 5, 6, 7, 9 and 10 of Ceplene/IL-2 therapy, corresponding to approximately every 3 months during this immunotherapy.
Pharmacodynamic effects of Ceplene plus low dose IL-2 (Ceplene/IL-2) by monitoring T and NK cell phenotypes and their functionality after the first and third cycles of treatment | Baseline vs Cycle 1 and 3
  The quantitative and qualitative pharmacodynamic effects of Ceplene/IL-2 on the immune responses of T and NK cells will be assessed as follows:
  1. Changes in T and NK cell phenotypes (CD56, CD3, CD4, CD8) in peripheral blood from Day 1 (baseline) to Day 21‡ of Cycle 1 and from Day 1 (pre-treatment Cycle 3) to Day 21‡ of Cycle 3.
  2. Changes in immune response markers (CD3, NKp46 [and other NCRs], CD25, CD69, and IFN-γ) in peripheral blood from Day 1 (baseline) to Day 21‡ of Cycle 1 and from Day 1 (pre-treatment Cycle 3) to Day 21‡ of Cycle 3

SECONDARY OUTCOMES:
Duration of LFS | up to 2 years
  Duration of LFS: LFS will be defined as the time from achieving CR after successful induction therapy until relapse of AML (defined as 5% or more blast cells in the bone marrow).

CONTACTS AND LOCATIONS:
Overall Officials: Robin FOA, MD, PhD, Study Chair — Università degli Studi di Roma "La Sapienza" Dipartimento di Biotecnologie Cellulari ed Ematolgia; Mats L Brune, MD, PhD, Principal Investigator — Sahlgrenska Academy University of Gothenburg, Gothenburg, Sweden
Locations (1):
- Sahlgrenska Academy, University of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Derived] Hussein BA, Hallner A, Wennstrom L, Brune M, Martner A, Hellstrand K, Bernson E, Thoren FB. Impact of NK Cell Activating Receptor Gene Variants on Receptor Expression and Outcome of Immunotherapy in Acute Myeloid Leukemia. Front Immunol. 2021 Dec 9;12:796072. doi: 10.3389/fimmu.2021.796072. eCollection 2021. PMID 34956230
- [Derived] Grauers Wiktorin H, Aydin E, Christenson K, Issdisai N, Thoren FB, Hellstrand K, Martner A. Impact of IL-1beta and the IL-1R antagonist on relapse risk and survival in AML patients undergoing immunotherapy for remission maintenance. Oncoimmunology. 2021 Jul 25;10(1):1944538. doi: 10.1080/2162402X.2021.1944538. eCollection 2021. PMID 34367728
- [Derived] Grauers Wiktorin H, Nilsson MS, Kiffin R, Sander FE, Lenox B, Rydstrom A, Hellstrand K, Martner A. Histamine targets myeloid-derived suppressor cells and improves the anti-tumor efficacy of PD-1/PD-L1 checkpoint blockade. Cancer Immunol Immunother. 2019 Feb;68(2):163-174. doi: 10.1007/s00262-018-2253-6. Epub 2018 Oct 12. PMID 30315349
- [Derived] Sander FE, Nilsson M, Rydstrom A, Aurelius J, Riise RE, Movitz C, Bernson E, Kiffin R, Stahlberg A, Brune M, Foa R, Hellstrand K, Thoren FB, Martner A. Role of regulatory T cells in acute myeloid leukemia patients undergoing relapse-preventive immunotherapy. Cancer Immunol Immunother. 2017 Nov;66(11):1473-1484. doi: 10.1007/s00262-017-2040-9. Epub 2017 Jul 18. PMID 28721449
- [Derived] Bernson E, Hallner A, Sander FE, Wilsson O, Werlenius O, Rydstrom A, Kiffin R, Brune M, Foa R, Aurelius J, Martner A, Hellstrand K, Thoren FB. Impact of killer-immunoglobulin-like receptor and human leukocyte antigen genotypes on the efficacy of immunotherapy in acute myeloid leukemia. Leukemia. 2017 Dec;31(12):2552-2559. doi: 10.1038/leu.2017.151. Epub 2017 May 22. PMID 28529313
- [Derived] Rydstrom A, Hallner A, Aurelius J, Sander FE, Bernson E, Kiffin R, Thoren FB, Hellstrand K, Martner A. Dynamics of myeloid cell populations during relapse-preventive immunotherapy in acute myeloid leukemia. J Leukoc Biol. 2017 Aug;102(2):467-474. doi: 10.1189/jlb.5VMA1116-455R. Epub 2017 Feb 24. PMID 28235771
- [Derived] Sander FE, Rydstrom A, Bernson E, Kiffin R, Riise R, Aurelius J, Anderson H, Brune M, Foa R, Hellstrand K, Thoren FB, Martner A. Dynamics of cytotoxic T cell subsets during immunotherapy predicts outcome in acute myeloid leukemia. Oncotarget. 2016 Feb 16;7(7):7586-96. doi: 10.18632/oncotarget.7210. PMID 26863635